CLINICAL TRIAL: NCT00030901
Title: L-Selenium-Based Chemoprevention Of Prostate Cancer Among Men With High Grade Prostatic Intraepithelial Neoplasia
Brief Title: S9917, Selenium in Preventing Cancer in Patients With Neoplasia of the Prostate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CDR0000069210; U10CA037429 (NIH); S9917 (Other: SWOG); CALGB-70004 (Other: CALGB); NCI-P02-0203 (Other: NCI grant)
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Results first posted 2013-02-06 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-01

CONDITIONS: Precancerous/Nonmalignant Condition; Prostate Cancer
Keywords: prostate cancer; high grade prostatic intraepithelial neoplasia
MeSH Terms: conditions — Precancerous Conditions; Prostatic Neoplasms | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-selenomethionine (Active Comparator): L-selenomethionine (Selenium)one tablet by mouth daily for 3 years.
  Interventions: Drug: L-selenomethionine
- L-selenomethionine placebo (Placebo Comparator): L-selenomethionine placebo one tablet by mouth daily for 3 years
  Interventions: Drug: L-selenomethionine placebo

INTERVENTIONS:
Drug: L-selenomethionine — Randomization between active L-selenomethionine and placebo
  Other Names: Selenium
  Arms: L-selenomethionine
Drug: L-selenomethionine placebo — Randomization between active L-selenomethionine and placebo
  Other Names: placebo
  Arms: L-selenomethionine placebo

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development of cancer. The use of selenium may be an effective way to prevent prostate cancer in patients who have neoplasia of the prostate.

PURPOSE: Randomized phase III trial to study the effectiveness of selenium in preventing prostate cancer in patients who have neoplasia of the prostate.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effects of selenium versus placebo on the 3-year incidence rate of prostate cancer in patients with high-grade prostatic intraepithelial neoplasia.
* Compare the toxicity of these regimens in these patients.
* Compare the effects of these regimens on the rate of increase in prostate-specific antigen (PSA) in these patients.
* Compare the effects of these regimens on prostatic cellular proliferation and apoptosis, degradation of basal cell integrity of prostatic ducts, and changes in nuclear chromatin patterns in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to age (40-60 vs 61 and over), race (African American vs other), baseline PSA (less than 4 ng/mL vs 4-10 ng/mL), concurrent vitamin E supplementation (yes vs no), and cores obtained from initial biopsy (10 or more vs less than 10). Patients are randomized to 1 of 2 arms.

* Arm I: Patients receive oral selenium once daily.
* Arm II: Patients receive oral placebo once daily. Treatment in both arms continues for 3 years in the absence of progression to prostate cancer or unacceptable toxicity.

Patients are followed every 6 months for 2 years and then annually for 8 years.

PROJECTED ACCRUAL: A total of 465 patients will be randomized for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of high-grade prostatic intraepithelial neoplasia with no evidence of cancer

  * Documented by a digital rectal exam and biopsy of the prostate with transrectal ultrasound guidance (required if fewer than 6 cores obtained in biopsy) meeting one of the following conditions:

    * Biopsy yielded fewer than 10 cores within the past 24 months OR yielded more than 10 cores 6-24 months before study
    * Biopsy yielded 10 or more cores within the past 6 months
* PSA ≤ 10 ng/mL (≤ 5 ng/mL for patients who have received finasteride or other androgen suppressor within the past 2 months)
* American Urological Association symptom score of less than 20

PATIENT CHARACTERISTICS:

Age:

* 40 and over

Performance status:

* SWOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or adequately treated stage I or II cancer that is in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* See Disease Characteristics
* No concurrent finasteride or any other androgen suppressor

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 30 days since prior daily dietary supplements containing 50 micrograms or more of selenium
* No concurrent daily dietary supplements containing more than 50 micrograms of selenium

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2000-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Marshall, PhD, Study Chair — Roswell Park Cancer Institute; David Jarrard, MD, Study Chair — University of Wisconsin, Madison; W. Robert Lee, MD, Study Chair — Wake Forest University Health Sciences

REFERENCES:
- [Result] Marshall JR, Sakr W, Wood D, Berry D, Tangen C, Parker F, Thompson I, Lippman SM, Lieberman R, Alberts D, Jarrard D, Coltman C, Greenwald P, Minasian L, Crawford ED. Design and progress of a trial of selenium to prevent prostate cancer among men with high-grade prostatic intraepithelial neoplasia. Cancer Epidemiol Biomarkers Prev. 2006 Aug;15(8):1479-84. doi: 10.1158/1055-9965.EPI-05-0585. PMID 16896036
- [Result] Sakr WA, Faulkner JR, Wood D: Low rate of confirming prostate cancer on repeat biopsies following diagnosis of high grade prostatic intraepithelial neoplasia: preliminary analysis of Southwest Oncology Group study s9917. [Abstract] Proceedings of the American Association for Cancer Research 45: A-1333, 305, 2004.

RESULTS

PARTICIPANT FLOW:
Groups:
- Selenium: Patients receive oral selenium once daily for 3 years
- Placebo: Patients receive oral placebo once daily for 3 years
Period: Initial Registration
Arm/Group | All Patients | Selenium | Placebo
Started | 619 | 0 | 0
Completed | 452 | 0 | 0
Not Completed | 167 | 0 | 0
Not completed — Ineligible | 167 | 0 | 0
Period: Randomization
Arm/Group | All Patients | Selenium | Placebo
Started | 0 | 227 | 225
Eligible | 0 | 212 | 211
Completed | 0 | 126 | 137
Not Completed | 0 | 101 | 88
Not completed — Adverse Event | 0 | 11 | 7
Not completed — Refusal Unrelated to Adverse Event | 0 | 16 | 10
Not completed — Progression/Relapse | 0 | 22 | 21
Not completed — Death | 0 | 1 | 3
Not completed — Other | 0 | 36 | 33
Not completed — Ineligible | 0 | 15 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Selenium | Placebo | Total
Number analyzed (Participants) | 212 | 211 | 423
Age Continuous [Median (Full Range); unit: years] | 65.90 [42.2 to 80.10] | 65.30 [44.9 to 82.7] | 65.65 [42.2 to 82.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 212 | 211 | 423
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 13 | 17
  Not Hispanic or Latino | 195 | 187 | 382
  Unknown or Not Reported | 13 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 26 | 26 | 52
  White | 180 | 173 | 353
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 6 | 6
Age [Number; unit: participants]
  <50 years | 9 | 7 | 16
  50-54 years | 20 | 20 | 40
  55-60 years | 28 | 35 | 63
  61-70 years | 96 | 98 | 194
  >70 years | 59 | 51 | 110
Baseline Prostate-Specific Antigen (PSA) - reported by site [Number; unit: participants]
  <4 ng/mL | 81 | 90 | 171
  4-10 ng/mL | 131 | 121 | 252

OUTCOME MEASURES:

1. Primary Outcome: Presence of Carcinoma of the Prostate as Measured by Biopsy
Description: The primary endpoint is biopsy-proven presence/absence of carcinoma of the prostate within 3 years after randomization to treatment. An end-of-study biopsy at 3 years after randomization will be used to determine presence/absence of prostate carcinoma in those patients not previously diagnosed with prostate carcinoma on study. Biopsies performed within ± 90 days of the 3-year anniversary will be considered end-of-study biopsies. Pathologically confirmed presence of prostate carcinoma may be determined at any time during the 3 years and 90 days after randomization, but absence can only be determined by the end-of-study biopsy.
Time Frame: 3 years
Population: All eligible randomized patients who started treatment and have prostate cancer known through an interim biopsy or a biopsy taken at +/- 90 days of the end of study were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Selenium | Placebo
Number analyzed (Participants) | 135 | 134
participants | 48 | 49
Statistical Analysis 1: Comparison: Selenium vs Placebo; With target sample size of 466 randomized patients (233 per arm), there is a 90% of power to detect a one-third reduction in the three-year incidence rate of prostate cancer. The alpha level is set at 0.025, one-sided; Test type: Superiority or Other; p = 0.73, Regression, Logistic — P-value is adjusted for stratification factors age older than 60, African American, baseline PSA, and vitamin E supplementation

2. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 2.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: 3 months after randomization and then every 3 months for 3 years
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | Selenium | Placebo
Number analyzed (Participants) | 203 | 202
Participants
  Cardiac ischemia/infarction | 0 | 1
  GI-other | 0 | 1
  Rash/desquamation | 1 | 0
  Urinary frequency/urgency | 0 | 1

ADVERSE EVENTS:
Time Frame: 3 months after randomization and then every 3 months for 3 years
Arm/Group | Selenium | Placebo
Serious Adverse Events (participants affected / at risk) | 9/203 | 4/202
Other Adverse Events (participants affected / at risk) | 54/203 | 57/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selenium (N=203) | Placebo (N=202)
Cardiac ischemia/infarction (Cardiac disorders) | 2 | 1
Cardiovascular-other (Cardiac disorders) | 2 | 1
LVEF decrease/CHF (Cardiac disorders) | 1 | 0
Supraventricular arrhythmia (Cardiac disorders) | 1 | 0
Abdominal pain/cramping (Gastrointestinal disorders) | 1 | 0
GI-other (Gastrointestinal disorders) | 1 | 0
Reportable adverse event, NOS (General disorders) | 0 | 1
Cerebrovascular ischemia (Nervous system disorders) | 1 | 0
Neuro-other (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusions (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombosis/embolism (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Selenium (N=203) | Placebo (N=202)
GI-other (Gastrointestinal disorders) | 13 | 11
Fatigue/malaise/lethargy (General disorders) | 28 | 18
Urinary frequency/urgency (Renal and urinary disorders) | 17 | 23
Nail changes (Skin and subcutaneous tissue disorders) | 16 | 11
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No